CLINICAL TRIAL: NCT00366821
Title: Retrospective Review of the Outcomes of Newborns With Genetic Abnormalities
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 06-141
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Congenital Disorders
Keywords: cardiac; pediatric; genetic
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Examine the outcomes following cardiac surgery in those newborns with genetic abnormalities.
- 2: Examine the outcomes following cardiac surgery in newborns without genetic abnormalities.

SUMMARY:
Our hope is that the information from this retrospective study will provide information to better serve our patients and their parents with risk stratification (levels of risk) and clinical expectations of patients after cardiac surgery who have genetic abnormalities and those who do not have genetic abnormalities.

DETAILED DESCRIPTION:
Screening for genetic/chromosomal abnormalities has become more frequent both pre-natally and post-natally. Therefore, we plan to review the outcomes in newborns with genetic abnormalities after cardiac surgery compared to those newborns without genetic abnormalities after cardiac surgery.

We wish to examine the outcomes following cardiac surgery in newborns with genetic abnormalities compared to those newborns without genetic abnormalities. We will compare morality rates and co-morbidities in each group.

We will retrospectively review the cardiac surgical database and patient medical records for all neonates (newborns < 30 days of age) who underwent cardiac surgery from January 1, 2002 through May 31, 2006 at Children's Healthcare of Atlanta. We plan to collect data on approximately 1000 patients including date of birth, age, weight, gestation, prenatal diagnosis, genetic abnormality, cardiac defect, surgery, operative details, pre-op and post-op complications, length of time on ventilator, hospital stay and mortality for these patients.

We will review the patient outcome data available after their initial surgery through May 31, 2006. No patients will be contacted.

ELIGIBILITY:
Inclusion Criteria:

* neonates (newborns< 30 days of age)
* cardiac surgery between 1/1/02 - 5/31/06
* at Children's Healthcare of Atlanta

Exclusion Criteria:

* those who do not meet inclusion criteria

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients' charts will be reviewed from Children's Healtcare of Atlanta between January 1, 2002 through December 31, 2006 of all neonates who underwent cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2002-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
We wish to examine the outcomes following cardiac surgery in newborns with genetic abnormalities compared to those newborns without genetic abnormalities. | 5 years
  We wish to examine the outcomes following cardiac surgery in newborns with genetic abnormalities compared to those newborns without genetic abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Simsic, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States